CLINICAL TRIAL: NCT02205463
Title: A Phase Ib Study of KD019 Plus Trastuzumab in Patients With HER2 Overexpressed or Amplified Metastatic or Unresectable Adenocarcinoma of Esophagus, Gastroesophageal Junction and Stomach
Brief Title: KD019 and Trastuzumab in Patients With Esophagus, Gastroesophageal Junction and Stomach Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: IND application withdrawn
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s14-01171
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Esophageal Cancer; Stomach Cancer
Keywords: Esophagus; Gastroesophageal Junction; Stomach; Gastric; Cancer; HER2; Metastatic; Adenocarcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Neoplasms; Neoplasm Metastasis; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KD019 (Experimental): Patients with HER2+ metastatic or unresectable adenocarcinoma of the esophagus, gastroesophageal junction or stomach will receive trastuzumab and mFOLFOX-6 in combination with KD019 to evaluate the safety, toxicity and MTD of this regimen. There will be four dose cohorts for KD019. KD019 will be administered orally continuously daily on a 28 day cycle. Trastuzumab and mFOLFOX-6 will be administered as infusions every 2 weeks at standard doses without escalation. The sequence on the days when all agents are administered will be KD019 followed by trastuzumab and mFOLFOX-6.
  Interventions: Drug: KD019

INTERVENTIONS:
Drug: KD019

SUMMARY:
This dose-escalation study is to determine the safety, maximum tolerated dose (MTD) and efficacy of KD019 in combination with trastuzumab and mFOLFOX-6.

DETAILED DESCRIPTION:
This is an open-label, single-arm, dose-escalation phase Ib study to determine the safety, maximum tolerated dose (MTD) and efficacy of KD019, a multi kinase inhibitor of EGFR, HER2, Src and VEGFR2, in combination with trastuzumab and mFOLFOX-6 for patients with human epidermal growth factor receptor 2 positive (HER2+) metastatic or unresectable adenocarcinoma of esophagus, gastroesophageal junction or stomach.

Patients with HER2+ metastatic or unresectable adenocarcinoma of the esophagus, gastroesophageal junction or stomach will receive trastuzumab and mFOLFOX-6 in combination with KD019 to evaluate the safety, toxicity and maximum tolerated dose of this regimen. There will be four dose cohorts for KD019. KD019 will be administered orally continuously daily on a 28 day cycle. Trastuzumab and mFOLFOX-6 will be administered as infusions every 2 weeks at standard doses without escalation. The sequence on the days when all agents are administered will be KD019 followed by trastuzumab and mFOLFOX-6.

Hypothesis A) KD019, a small molecule inhibitor of multiple receptor tyrosine kinases including EGFR, HER2, VEGFR-2 and Src, can be safely added, in an effective dose, to the every 2 week schedule of mFOLFOX-6 + trastuzumab for patients with metastatic or unresectable HER2+ adenocarcinoma of esophagus, GEJ or stomach

B) When added to mFOLFOX-6 + trastuzumab, KD019will increase response duration, progression free survival

Primary objective:

To assess the safety, tolerability, maximum tolerated dose (MTD), recommended phase II dosing (RP2D) of KD019 in combination of trastuzumab and mFOLFOX-6

Secondary objectives:

1. To characterize the pharmacokinetics (PK) parameters of KD019 administered once daily in combination with every 2 week mFOLFOX-6 and trastuzumab in subjects with metastatic or unresectable HER2+ adenocarcinoma of the esophagus, gastroesophageal junction (GEJ) and stomach.
2. To evaluate tumor biopsy specimens pre- and post- treatment with KD019 and trastuzumab for changes in target receptors and correlate with response

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

* Pathologically confirmed diagnosis of adenocarcinoma of stomach, GEJ or esophagus (central confirmation is not required). Primary tumor or metastatic lesion must be HER2+ documented as HER2 gene amplification by FISH as positive (HER2:CEP17 ratio of ≥2.0) or IHC 3+.
* Metastatic or unresectable adenocarcinoma of stomach, GEJ, or esophagus that is evaluable or that is measurable for response as per RECIST 1.1 criteria, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral computed tomography (CT) scan.
* Adult subjects greater than 18 years of age
* Patients who received postoperative adjuvant therapy with a single-agent fluoropyrimidine and radiation are eligible.
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1.
* Adequate organ and bone marrow functions defined as follows:

oAbsolute neutrophil count >1,500 cells/ul

* Platelets >100,000/ul
* Hemoglobin >9.0g/dl
* INR < or equal to 1.5 or INR < or equal to 3 if patient is on warfarin
* Serum creatinine < or equal to 1.5 times upper limit of normal (ULN) or calculated creatinine clearance (CRCL) > or equal to 60ml/min
* Serum electrolytes within the normal range (per institution standard) during screening.
* Total bilirubin less than or equal to 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < or equal to 3 times ULN
* Albumin > or equal to 3g/dL

  * No history of another malignancy in the past 5 years, except treated non-melanoma skin cancer or superficial bladder cancer or carcinoma-in-situ of the cervix
  * No coexisting medical problems of sufficient severity to limit compliance with the study
  * Ability to understand and sign a written informed consent document. Patient must have willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
  * Female subjects of childbearing potential must have a negative serum pregnancy test prior to study entry (positive urine tests are to be confirmed by serum test).
  * Female subjects of childbearing potential and males must agree to use a highly effective method of contraception (<1% per year failure rate) for the duration of study treatment and for six months after discontinuation of the study drug. Highly effective birth control methods include implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence, or vasectomy for males.

Exclusion Criteria:

* Prior treatment chemotherapy or HER2-directed therapy for metastatic gastric, GEJ or esophageal adenocarcinoma chemotherapy.
* Prior peri-operative therapy with a platinum-containing regimen.
* Angina secondary to fluoropyrimidine therapy in the adjuvant setting
* Surgery, radiotherapy, or lesion ablative procedure to the only area of measurable/evaluable disease.
* Major surgery within 4 weeks prior to the first dose of KD019
* Left ventricular ejection fraction (EF) <50% at baseline as measured by multi-gated acquisition (MUGA) scan or echocardiogram (ECHO).
* Treatment with chronic immunosuppressants (e.g. cyclosporine following transplantation)
* Current known active infection with HIV, hepatitis B or C viruses
* Uncontrolled systemic disease
* Brain metastases that are:

  * Untreated or
  * Progressive or
  * Have required any type of therapy (including radiation, surgery, steroids or anticonvulsant therapy) to control symptoms from brain metastases within 60 days prior to the first study treatment
  * Leptomeningeal
  * Hemorrhagic
* Subject has evidence of pre-existing idiopathic pulmonary fibrosis on CT scan at baseline
* History of an invasive secondary primary malignancy diagnosed within the previous 3 years, except for appropriately treated stage I endometrial or cervical carcinoma, prostate carcinoma treated surgically or non-melanoma skin cancer.
* No other non-protocol antineoplastic agents will be permitted during this study
* Patients may not be receiving any other investigational agents.
* Women who are pregnant or lactating.
* Subject has any of the following EKG criteria:

  * Corrected QT interval (QTc) of >0.47 seconds
  * Finding of a left bundle branch block or right bundle bunch block
* Bradycardia defined as a heart rate of <50 beats per minute (bpm)
* Presence of a pacemaker or implantable cardioverter defibrillator (ICD)
* History of sustained ventricular arrhythmias (subjects with a history of atrial arrhythmias should be discussed with the sponsor before entry into the study)
* Family history of congenital long QT syndrome or unexplained sudden death.
* Moderate or severe pulmonary dysfunction
* History of clinically significant cardiac dysfunction including:

  * Unstable angina
  * History of myocardial infarction (MI) within 6 months prior to first study treatment
  * History of symptomatic CHF (grade >3 by NCI CTCAE or Class >II by New York Heart Association (NYHA) criteria or serious cardiac arrhythmia requiring treatment, with the exception of atrial fibrillation and paroxysmal supraventricular tachycardia
  * Uncontrolled hypertension defined as systolic blood pressure (SBP) ≥ 160 and/or diastolic blood pressure (DBP) ≥ 100 despite maximal medical therapy.
* Subject requires treatment with drugs known to be associated with torsades de pointes or significant QT interval prolongation.

  * Patients will be eligible for the study if they discontinue any medications listed in one week prior to registration and study enrollment.
  * Stable regimen of antidepressants of the SSRI class is allowed (common SSRIs include escitalopram oxalate, citalopram, fluvoxamine, paroxetine, sertraline and fluoxetine)
* Use of cytochrome P450 enzyme-inducing anti-epileptic drugs (such as phenytoin, carbamazepine or phenobarbital) is not allowed.
* Subject has a serum potassium or magnesium level outside the normal range despite repletion.
* Has gastrointestinal tract disease resulting in an inability to take or absorb oral medication.
* Inclusion or exclusion of patients on other medications, or severe acute/chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results will be at the judgment of the study investigator.
* Subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 Days
  To determine maximum tolerated dose (MTD) and RP2D of KD019 in combination with trastuzumab and mFOLFOX-6 when given to patients with HER2+ metastatic or unresectable adenocarcinoma of the esophagus, GEJ or stomach (gastric).

SECONDARY OUTCOMES:
Progression-Free Survival | 3 Years
  Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Tumor assessments will be performed using RECIST criteria (Version 1.1). Imaging scans may be done within 4 weeks prior to the first dose of study drug (baseline) and then every 12 weeks (±7 days) after the first dose of study drug until documented progression. Responses will be confirmed by repeat assessments between 28 and 35 days after the response criteria are first met.
Objective Response Rate | 3 Years
  Overall response rates are defined as partial response plus complete response. Tumor response will be based on Response evaluation Criteria in Solid Tumors (RECIST 1.1). Response rates will be estimated with exact 95% confidence intervals for each dose level. Kaplan Meier curves will be used to summarize progression free survival.
Duration of Response | 3 Years
  The duration of overall response is measured from the time measurement are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Tumor response will be based on Response evaluation Criteria in Solid Tumors (RECIST 1.1).
Clinical Benefit Rate | 3 Years
  Clinical benefit rate is defined as complete response plus partial response plus stable disease >16 weeks, and will be summarized descriptively. Tumor response will be based on Response evaluation Criteria in Solid Tumors (RECIST 1.1).
Pharmacokinetics of KD019 | Multiple
  Patients will undergo pharmacokinetics at the following time points:
  * Pre- 15 minutes pre-dosing: C1 D1, C1 D15 and then D1 only starting cycle 2 and thereafter Up to and including the cycle 6 visit.
  * Post- at 1 hour, 2 hours, and 4-6 hours post dosing: C1 D1, C1 D15 and 4-6 hours post dosing only on D1 only starting cycle 2 .
  * A PK sample will also be drawn if QTc(f) interval increases to an absolute value of >500 msec. The concentration of KD019 in these samples will be used to confirm exposure to KD019 and to further characterize the plasma PK of KD019 in this subject population.
  * 30 days post treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wu, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States